CLINICAL TRIAL: NCT01064557
Title: Guideline for the Treatment of Newly Diagnosed Patients Eith Acutypromyelocytic Leukemia, Aged > 12 Months (1 Year) and <75 Years, Using All-trans Retinoic Acid in Combination With Idarubicin
Brief Title: "AIDA" Protocol (LAP 0493)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIDA0493
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Leukemia
Keywords: Acute promyelocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: all-trans retinoic acid (ATRA)

SUMMARY:
The main purposes of the AIDA protocol are to test the role of intermittent maintenance therapy with ATRA, standard maintenance chemotherapy with methotrexate and 6-mercaptopurine of both in PCR negative patients at the end of the consolidation phase and to evaluate the role of allogeneic or autologous bone marrow transplantation in PCR positive patients at the end of the consolidation phase.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 months (1 year) and < 75 years
* Morphological newly diagnosis of APL
* Presence of the PML-RARa transcript
* No cardiac contraindications to anthracycline chemotherapy
* Serum creatinine <=2.5 mg/dL
* Serum alkaline phosphatase <= 3 times the normal upper limit
* Serum bilirubin <= 3 times the normal upper limit
* Serum SGOT <= 3 times the upper normal limit
* Negative pregnancy test
* Informed consent

Exclusion Criteria:

* Age <= 12 months and >=75 years
* absence of the PML-RARa transcript
* Pregnant of lactating women
* Presence of active serious infections that are not controlled by antibiotics
* Prior treatment with antileukemic therapy (excluded corticosteroids)
* Presence of severe concomitant psychiatric disease
* Presence of other concomitant malignant tumors, except basal cell carcinoma
* Concurrent treatment with cytotoxic chemotherapy or radiotherapy
* Cardiac contraindications to anthracycline chemotherapy
* Serum creatinine >2.5 mg/dL
* Serum alkaline phosphatase > 3 times the normal upper limit
* Serum bilirubin > 3 times the normal upper limit
* Serum SGOT > 3 times the upper normal limit
* Positive pregnancy test
* Absence of informed consent

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1068 (Estimated)
Dates: Start 1993-10; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To assess the role of maintenance therapy with ATRA, chemotherapy or both in PCR negative patients at the end of the consolidation phase.

SECONDARY OUTCOMES:
To assess the role of allogeneic or autologous bone marrow transplantation in PCR positive patients at the end of the consolidation phase
To evaluate the role of maintenance therapy with ATRA and chemotherapy in PCR positive patients at the end of the consolidation phase not eligible for a BMT procedure
To assess the efficacy, in terms of CR rate, and toxicity of an induction treatment combining ATRA with Idarubicin

CONTACTS AND LOCATIONS:
Locations (80):
- Department of Hematology - Middelheim Ziekenhuis, Antwerp, Belgium
- Department of Hematology - Klinikum Grosshadem - Ludwig Maxmilians, München, Germany
- Italy (75):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - Centro di Riferimento Oncologico, Aviano
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - ASL12 - Biella Ospedale degli Infermi - Dip. di Medicina e Geriatria - Struttura Complessa di Medicina Interna, Biella
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Comprensorio Sanitario di Bolzano - Azienda Sanitaria dell'Alto Adige - Ematologia e Centro TMO - Ospedale S.Maurizio, Bolzano
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Ferrara
  - Policlinico di Careggi, Università delgi studi di Firenze, Florence
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Ospedale S. Antonio Abate, Gallarate
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - Clinica Medica III - Padiglione 3 - Azienda Ospedale Università San Martino, Genova
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - Ospedale San Martino, Genova
  - Università degli Studi, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Divisione Ospedale Maggiore, Lodi
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera "S.Gerardo", Monza
  - A.S.L. Napoli 1 Ospedale San Giovanni Bosco, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - Servizio Sanitario Nazionale - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Struttura Complessa di Ematologia - Div. TERE- 4° piano - Padiglione Palermo, Napoli
  - Divisione di Oncologia Medica Ospedale Pierfortunato Calvi, Noale
  - Sez. di Ematologia Clinica Ospedale San Francesco, Nuoro
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Ospedale Cervello, Palermo
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Med. Int. ed Oncologia Medica IRCCS Policlinico S. Matteo, Pavia
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - Sezione di Medicina Interna e Scienze e Oncologiche (MISO ) Osp. S.Maria della Misericordia, Perugia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Unità operativa Medicina II Az. Osp. S. M. degli Angeli, Pordenone
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - A.O Umberto I, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Pr. Lo Coco, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, S. G. Rotondo
  - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Azienda Ospedaliera della Valtellina e della Valchiavenna, Sondalo
  - U.O.C. di Ematolgia - A.O. " SS Annunziata" - P.O. S.G. Moscati, Taranto
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza
- Netherlands (2):
  - Department of Hematology - Medical Center - Leiden University, Leiden
  - Department of Hematology - St Radboud University - Hospital, Nijmegen
- Department of Hematology - Ankara University School of Medicine - Ibni Sina Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Avvisati G, Lo Coco F, Diverio D, Falda M, Ferrara F, Lazzarino M, Russo D, Petti MC, Mandelli F. AIDA (all-trans retinoic acid + idarubicin) in newly diagnosed acute promyelocytic leukemia: a Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto (GIMEMA) pilot study. Blood. 1996 Aug 15;88(4):1390-8. PMID 8695858
- [Result] Avvisati G, Lo-Coco F, Paoloni FP, Petti MC, Diverio D, Vignetti M, Latagliata R, Specchia G, Baccarani M, Di Bona E, Fioritoni G, Marmont F, Rambaldi A, Di Raimondo F, Kropp MG, Pizzolo G, Pogliani EM, Rossi G, Cantore N, Nobile F, Gabbas A, Ferrara F, Fazi P, Amadori S, Mandelli F; GIMEMA, AIEOP, and EORTC Cooperative Groups. AIDA 0493 protocol for newly diagnosed acute promyelocytic leukemia: very long-term results and role of maintenance. Blood. 2011 May 5;117(18):4716-25. doi: 10.1182/blood-2010-08-302950. Epub 2011 Mar 8. PMID 21385856
- [Result] Latagliata R, Breccia M, Fazi P, Vignetti M, Di Raimondo F, Sborgia M, Vincelli D, Candoni A, Salvi F, Rupoli S, Martinelli G, Kropp MG, Tonso A, Venditti A, Melillo L, Cimino G, Petti MC, Avvisati G, Lo-Coco F, Mandelli F; GIMEMA Acute Leukaemia Working Party. GIMEMA AIDA 0493 amended protocol for elderly patients with acute promyelocytic leukaemia. Long-term results and prognostic factors. Br J Haematol. 2011 Sep;154(5):564-8. doi: 10.1111/j.1365-2141.2011.08593.x. Epub 2011 Jul 14. PMID 21751984
- See also: GIMEMA Foundation — http://www.gimema.it